CLINICAL TRIAL: NCT03639688
Title: The Ease of Threading the Endotracheal Tube Over the Fiberoptic Bronchoscope on the Left vs Right Lip Commissure
Brief Title: Endotracheal Tube Threading Over the Fiberoptic Bronchoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Marwan Rizk, Assistant Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANES.MR.02
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Fiberoptic Guided Intubation
Keywords: Endotracheal intubation; Fiberoptic bronchoscope

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left-sided threading (Placebo Comparator): Patients intubated with fiberoptic bronchoscope by threading the tube on the left labial commissure
  Interventions: Procedure: Threading on the left lip commissure
- Right-sided threading (Active Comparator): Patients intubated with fiberoptic bronchoscope by threading the tube on the right labial commissure
  Interventions: Procedure: Threading on the right lip commmissure

INTERVENTIONS:
Procedure: Threading on the left lip commissure — Threading of the endotracheal tube over the fiberoptic bronchscope from the left lip commissure
  Arms: Left-sided threading
Procedure: Threading on the right lip commmissure — Threading of the endotracheal tube over the fiberoptic bronchoscope from the right lip commissure
  Arms: Right-sided threading

SUMMARY:
The goal of this study is to assess the ease of ETT threading over the FOB on the right or left labial commissures in patients aging between 18 and 70 years old with ASA score I-II and undergoing any type of surgery. The main question it aims to answer is whether threading the tube on the right labial commissure during FOB intubation has a better success rate than threading the tube on the left labial commissure. Participants will be randomized via a computerized system into 2 groups (Group 1: Patients intubated with FOB by threading the tube on the left labial commissure and Group 2: Patients intubated with FOB by threading the tube on the right labial commissure). Researchers will compare the success rate of threading the tube on first trial, number of ETT threading trials, time to success, and incidence of intra-procedural complication between the two groups to see if threading the tube on the right labial commissure during FOB intubation has a better success rate than threading the tube on the left labial commissure.

DETAILED DESCRIPTION:
Fiberoptic bronchoscope (FOB) intubation is the gold standard technique for intubating patients with predicted difficult airway. Different maneuvers have been used to facilitate threading the endotracheal tube (ETT) over the fiberoptic bronchoscope including jaw thrust, stretching the tongue, rotating the ETT 90 degrees anticlockwise or using smaller tubes. To our knowledge threading the ETT with the FOB on the left or right lip commissures has not been investigated previously. Improving the ease of ETT threading on the right or left labial commissures could change our FOB intubation management.

The aim is to assess the ease of ETT threading over the FOB on the right or left labial commissures.

Patients between 18 and 70 years old with ASA score I-II and undergoing any type of surgery in the operating rooms at the American University of Beirut Medical Center will be randomized via a computerized system into 2 groups:

Group 1: Patients intubated with FOB by threading the tube on the left labial commissure Group 2: Patients intubated with FOB by threading the tube on the right labial commissure The primary outcome is the success rate of threading the tube on first trial. Secondary outcomes include number of ETT threading trials, time to success, and incidence of intra-procedural complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 70 years
* Any surgery requiring general anesthesia
* ASA 1 and 2

Exclusion Criteria:

* Patients aged less than 18 or more than 70 years old.
* ASA 3 and 4 patients.
* Patients who need a rapid sequence induction (including pregnant women) or those who have an increased risk of aspiration.
* Patients who need awake fiberoptic intubation for a difficult airway or any other reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
success rate of intubation | up to 30 minutes from anesthesia initiation
  the success rate of intubation after threading the tube on the designated commissure on the first trial

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Rizk, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon